CLINICAL TRIAL: NCT01682161
Title: An Open-Label, Comparative Study of Immediate or Delayed Switch to Paliperidone Palmitate in Patients Unsatisfied With Current Oral Atypical Antipsychotics to Evaluate the Evolution of Medication Satisfaction and Adherence
Brief Title: A Comparative Study to Evaluate the Evolution of Medication Satisfaction and Adherence in Patients Unsatisfied With Current Oral Atypical Antipsychotics by Switching Medication to Paliperidone Palmitate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100740; R092670SCH4010 (Other: Janssen Korea, Ltd., Korea); PALM-KOR-4001 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Palmitate; Invega Sustenna; Antipsychotics; Atypical antipsychotics; Medication Satisfaction and Adherence
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Immediate switch) (Experimental): Paliperidone palmitate will be administered immediately after randomization and will be continued throughout the treatment phase.
  Interventions: Drug: Paliperidone palmitate
- Group 2 (Delayed switch) (Experimental): Current oral antipsychotics will be continued until Week 8, and later on paliperidone palmitate will be administered.
  Interventions: Drug: Paliperidone palmitate

INTERVENTIONS:
Drug: Paliperidone palmitate — Paliperidone palmitate will be administrated in accordance with each product's information. Recommended initial loading doses are 150 mg equivalent on Day 1 and 100 mg equivalent on Day 8, followed by subsequent once-monthly administration with 75 mg equivalent or flexible dose between 25 mg and 150 mg equivalent.
  Other Names: INVEGA SUSTENNA

SUMMARY:
The purpose of this study is to evaluate the change of medication satisfaction measured by Medication Satisfaction Questionnaire (MSQ) from baseline to endpoint for patients who are switched into paliperidone palmitate, either immediately or in a delayed mode.

DETAILED DESCRIPTION:
This is a prospective (patients are first identified and then followed forward as time passes), multicenter (study conducted at multiple sites), randomized (the study medication is assigned by chance), comparative and open-labeled (all people know the identity of the intervention) study.

The study mainly consists of 3 phases including, the screening phase (14 days before administration of study medication), treatment phase, and the follow-up phase (28 days after the last dose of the study medication). In the treatment phase, patients will be randomly assigned equally in 2 groups (Group 1 and Group 2), on the basis of known and unknown characteristics. Group 1 (immediate switch group): Patients will be administered with paliperidone palmitate immediately after randomization and will continue throughout the treatment phase. Group 2 (delayed switch group): Patients will remain on current oral antipsychotics until Week 8, and later on will be completely switched to paliperidone palmitate. However, during the first 8 weeks if the symptoms or satisfaction with MSQ further deteriorates for Group 2, they may be switched into paliperidone palmitate earlier.

Safety evaluations will include evaluation of adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination and these will be monitored throughout the study.

The total duration of the study will be approximately 148 days.

ELIGIBILITY:
Inclusion Criteria:- Meet diagnostic criteria for schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders Version IV

* Dissatisfied with current medication (Medication Satisfaction Questionnaire score of less than or equal to 4) or by clinician's judgment and who may benefit from switching medication
* Have received an oral antipsychotic for at least 4 weeks before randomization
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

History of neuroleptic malignant syndrome

* Presence of congenital prolongation of the QT interval - History of treatment with depot antipsychotics, including long-acting injectable risperidone and paliperidone palmitate, within 90 days of the screening visit; or any treatment with clozapine within the previous 60 days
* Any relevant medical history or current presence of systemic disease
* Significant risk of suicidal, homicidal or violent ideation or behavior as clinically assessed by the investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 21 in scores of Medication Satisfaction Questionnaire (MSQ) | Screening (Week -2), baseline (Week 0), Week 1, Week 5, Week 8, Week 9, Week 13, Week 17, and Week 21
  MSQ is designed to assess treatment satisfaction among patients with schizophrenia. The responses will be assessed on a 7-point Likert-type scale rated as follows: 1=extremely dissatisfied, 2=very dissatisfied, 3=somewhat dissatisfied, 4=neither satisfied nor dissatisfied, 5=somewhat satisfied, 6=very satisfied, and 7=extremely satisfied.

SECONDARY OUTCOMES:
Change from baseline to Week 21 in scores of Treatment Satisfaction Questionnaire for Medication (TSQM) | Screening, baseline, Week 1, Week 5, Week 8, Week 9, Week 13, Week 17, and Week 21
  The TSQM is a 14-item subject assessed evaluation of treatment medication using a 7-point Likert-type scale rated as follows: 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Somewhat Dissatisfied, 4=Neither Satisfied Nor Dissatisfied, 5=Somewhat Satisfied, 6=Very Satisfied, 7= Extremely Satisfied.
Change from baseline to Week 21 in scores of Positive and Negative Syndrome Scale (PANSS) | Baseline, Week 8, and Week 21
  The PANSS is a medical scale used for measuring symptom severity of patients with schizophrenia. The neuropsychiatric symptoms of schizophrenia will be assessed using the 30-item PANSS scale. Each item is rated as follows: 1=absent, 2=Minimal, 3=Mild, 4=Moderate, 5=Moderate Severe, 6=Severe, and 7=Extreme.
Change from baseline to Week 21 in scores of Clinical Global Impression - Severity (CGI-S) scale | Baseline, Week 1, Week 5, Week 8, Week 9, Week 13, Week 17, and Week 21
  The CGI-S rating scale is used to rate the severity of a patient's psychotic condition on a 7-point scale. It is rated as follows: 1=Normal, not at all ill, 2=Borderline mentally ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Among the most extremely ill.
Change from baseline to Week 21 in scores of Personal and Social Performance (PSP) scale | Baseline, Week 8, and Week 21
  The PSP is a clinician rated instrument providing an overall rating of personal and social functioning in patients with schizophrenia on a scale of 1-100. The scale defines a continuum from grossly impaired functioning, in which total lack of autonomy in basic functioning and survival risk is evident, to excellent functioning. Four domains of functioning are considered in the rating: 1) socially useful activities, including work and study, 2) personal and social relationships, 3) self-care, and 4) disturbing and aggressive behavior.
Score of Mediation Adherence Rating Scale (MARS) | Baseline
  The MARS is a 10-items self-rating scale to measure the adherence of the drug medication for psychosis. Each item is answered "yes/no" and the total score ranges from 0 points (Low medication adherence) to 10 points (High medication adherence).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (9):
- South Korea (9):
  - Buchun
  - Cheonan
  - Chungcheongbuk-Do
  - Daegu
  - Goyang
  - Gyeonggi-do
  - Incheon
  - Seognam-Si, Kyungki-Do
  - Seoul

REFERENCES:
- See also: An open-label, comparative study of immediate or delayed switch to paliperidone palmitate in patients unsatisfied with current oral atypical antipsychotics to evaluate the evolution of medication satisfaction and adherence — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3405&filename=CR100740_CSR.pdf